CLINICAL TRIAL: NCT02259231
Title: An Open-label, Multicenter, Dose-escalation, Phase 1b/2 Study of the Safety, Efficacy, Pharmacodynamics, and Pharmacokinetics of RTA 408 in Combination With Ipilimumab or Nivolumab in the Treatment of Patients With Unresectable or Metastatic Melanoma
Brief Title: RTA 408 Capsules in Patients With Melanoma - REVEAL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: RTA 408-C-1401
Record Dates: First submitted 2014-10-03; First posted 2014-10-08 (Estimated); Results first posted 2021-06-24 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Melanoma; Unresectable (Stage III) Melanoma; Metastatic (Stage IV) Melanoma
Keywords: RTA 408; RTA 408 Capsules; Myeloid-derived suppressor cells (MDSDs); iNOS; Melanoma; Checkpoint inhibitor; omaveloxolone
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — omaveloxolone; ORF 50 transactivator; Ipilimumab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Omaveloxolone 5 mg & ipilimumab (Experimental): Omaveloxolone (RTA 408) capsules, Dose1 taken orally once daily for 168 weeks, plus ipilimumab (3 mg/kg) administered at weeks 1, 4, 7, and 10.
  Interventions: Drug: Omaveloxolone Capsules (2.5 mg/capsule); Drug: Ipilimumab (3 mg/kg)
- Omaveloxolone 10 mg & ipilimumab (Experimental): Omaveloxolone (RTA 408) capsules, 10 mg taken orally once daily for 168 weeks, plus ipilimumab (3 mg/kg) administered at weeks 1, 4, 7, and 10.
  Interventions: Drug: Ipilimumab (3 mg/kg); Drug: Omaveloxolone Capsules (10 mg/capsule)
- Omaveloxolone 5 mg & nivolumab (Experimental): Omaveloxolone (RTA 408) capsules, 5 mg taken orally once daily for 168 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Interventions: Drug: Omaveloxolone Capsules (2.5 mg/capsule); Drug: Nivolumab (240 mg)
- Omaveloxolone 10 mg & nivolumab (Experimental): Omaveloxolone (RTA 408) capsules, 10 mg taken orally once daily for 168 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Interventions: Drug: Nivolumab (240 mg); Drug: Omaveloxolone Capsules (10 mg/capsule)
- Omaveloxolone 20 mg & nivolumab (Experimental): Omaveloxolone (RTA 408) capsules, 20 mg taken orally once daily for 168 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Interventions: Drug: Nivolumab (240 mg); Drug: Omaveloxolone Capsules (10 mg/capsule)
- Omaveloxolone 100 mg & nivolumab (Experimental): Omaveloxolone (RTA 408) capsules, 100 mg taken orally once daily for 168 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Interventions: Drug: Nivolumab (240 mg); Drug: Omaveloxolone Capsules (50 mg/capsule)
- Omaveloxolone 150 mg & nivolumab (Experimental): Omaveloxolone (RTA 408) capsules, 150 mg taken orally once daily for 168 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Interventions: Drug: Nivolumab (240 mg); Drug: Omaveloxolone Capsules (50 mg/capsule)

INTERVENTIONS:
Drug: Omaveloxolone Capsules (2.5 mg/capsule) — Capsules containing 2.5 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
  Other Names: RTA 408 Capsules (2.5 mg/capsule)
  Arms: Omaveloxolone 5 mg & ipilimumab; Omaveloxolone 5 mg & nivolumab
Drug: Ipilimumab (3 mg/kg) — Sterile solution containing ipilimumab to be delivered intravenously at 3mg/kg
  Other Names: Yervoy
  Arms: Omaveloxolone 10 mg & ipilimumab; Omaveloxolone 5 mg & ipilimumab
Drug: Nivolumab (240 mg) — Sterile solution containing nivolumab to be delivered intravenously at 240 mg
  Other Names: Opdivo
  Arms: Omaveloxolone 10 mg & nivolumab; Omaveloxolone 100 mg & nivolumab; Omaveloxolone 150 mg & nivolumab; Omaveloxolone 20 mg & nivolumab; Omaveloxolone 5 mg & nivolumab
Drug: Omaveloxolone Capsules (10 mg/capsule) — Capsules containing 10 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
  Other Names: RTA 408 Capsules (10 mg/capsule)
  Arms: Omaveloxolone 10 mg & ipilimumab; Omaveloxolone 10 mg & nivolumab; Omaveloxolone 20 mg & nivolumab
Drug: Omaveloxolone Capsules (50 mg/capsule) — Capsules containing 50 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
  Other Names: RTA 408 Capsules (50 mg/capsule)
  Arms: Omaveloxolone 100 mg & nivolumab; Omaveloxolone 150 mg & nivolumab

SUMMARY:
Malignant melanoma is a leading cause of death from cutaneous malignancies, accounting for approximately three-fourths of all skin cancer deaths. For metastatic or unresectable melanomas, standard treatment options include immune checkpoint inhibitors (e.g., ipilimumab and nivolumab) and other therapies, however, approved therapies are rarely curative.

It is now well accepted that tumors are able to evade detection and eradication by the immune system, even though many tumor types, particularly melanoma, are capable of eliciting a strong immune response (Swann, 2007). Substantial mechanistic work in recent years has revealed the key role of myeloid-derived suppressor cells (MDSCs) in masking cancer cells from the immune system, promoting both tumor progression and resistance to cancer immunotherapy. The immune-suppressive effect of MDSCs is dependent on the production of reactive oxygen species (ROS) and reactive nitrogen species (RNS). High levels of these reactive molecules and their by-products, such as nitrotyrosine, have been correlated with poor clinical outcomes in melanoma. Currently available melanoma therapies do not target MDSCs.

In animals, RTA 408 significantly reduces tumor nitrotyrosine burden, inhibits the activity of MDSCs, and augments T-cell anticancer activity at relevant doses. Thus, through inhibition of MDSC activity and suppression of tumor ROS/RNS, RTA 408 may work in combination with T-cell-activating therapeutics such as ipilimumab to enhance the natural immune anticancer response. RTA 408 also has direct anticancer effects via inhibition of NF-kappa B. Chronic activation of NF-kappa B is associated with tumor progression, metastasis, and resistance to therapy.

This proposed study is designed to assess the safety, efficacy, pharmacodynamics, and pharmacokinetics of omaveloxolone (RTA 408) in combination with ipilimumab or nivolumab in patients with unresectable or metastatic melanoma.

In this open-label, multicenter, dose-escalation, Phase 1b/2 study, patients who qualify will receive omaveloxolone (RTA 408) at the assigned dose level in combination with ipilimumab or nivolumab. Patients will receive omaveloxolone (RTA 408) orally once daily for 1 week prior to initiation of ipilimumab or nivolumab. For patients treated with ipilimumab , the run-in period will be followed by omaveloxolone (RTA 408) orally once daily in combination with ipilimumab administered at Weeks 1, 4, 7, and 10. After Week 10, patients will receive maintenance treatment with omaveloxolone (RTA 408) alone once daily. For patients treated with nivolumab, the run-in period will be followed by omaveloxolone (RTA 408) orally once daily in combination with nivolumab administered approximately every two weeks as clinically indicated. Each patient will continue at the assigned omaveloxolone (RTA 408) dose level until disease progression occurs, toxicity requiring discontinuation from study drug (i.e., RTA 408) is experienced, the patient has completed approximately 72 weeks of treatment, the patient is discontinued from the study drug for another reason, or the patient withdraws consent. Patients will return 4 weeks after omaveloxolone (RTA 408) treatment completion for a follow-up visit.

The starting omaveloxolone (RTA 408) dose level for the first dose-escalation cohort in this study has been selected based on available safety and pharmacodynamic data from a Phase 1 study of RTA 408 (NCT02029729). Subsequent cohorts will be enrolled at dose levels based on available safety and PD data from this study, but they will not be greater than 2-fold above the prior dose level.

Phase 1b (dose-escalation): In the phase 1b/2 portion of this study, 12 patients will be enrolled in each dose cohort, with six patients administered omaveloxolone (RTA 408) plus ipilimumab and the remaining six administered rTA 408 plus nivolumab. Subsequent cohorts will assess escalating the doses of omaveloxolone (RTA 408) administered in combination with ipilimumab or nivolumab. Dose escalation decisions will be based on ongoing review of all available safety information for enrolled patients.

Phase 2: The Phase 2 portion of the study may include separate expansion cohorts consisting of patients treated with either of the combination therapies. Each expansion cohort will include an additional 24 patients enrolled at the selected Phase 2 dose level to achieve a total of 30 patients at that omaveloxolone (RTA 408) dose in combination with ipilimumab or nivolumab.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years of age;
2. Have advanced, unresectable (Stage III) or metastatic (Stage IV) melanoma;
3. Be eligible for commercial receipt of therapy to be used in this study in combination with RTA 408 (i.e., ipilimumab or nivolumab in the Phase 1b portion and nivolumab only in the Phase 2 portion);
4. Have discontinued previous treatments for cancer;
5. Have discontinued previous experimental therapies and checkpoint inhibitor antibodies at least 28 days prior to the Randomization Visit

Exclusion Criteria:

1. Have received prior treatment with therapy to be used in this study in combination with RTA 408 (i.e., ipilimumab or nivolumab) if enrolling in the Phase 2 portion of the study. This criterion does not apply to patients enrolling in the Phase 1b portion of the study.
2. Have prior malignancy active within the previous 2 years;
3. Have any active autoimmune disease or a history of known or suspected autoimmune disease;
4. History of brain metastases that meet certain conditions;
5. History of specific cardiovascular abnormalities;
6. Have known active fungal, bacterial, and/or viral infection, including human immunodeficiency virus (HIV) or hepatitis virus (A,B, or C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-07-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Southern Cancer Center, Mobile, Alabama
  - Highlands Oncology Group, Fayetteville, Arkansas
  - University of Colorado Cancer Center, Anschutz Cancer Pavilion, Aurora, Colorado
  - Christiana Hospital Helen F. Graham Cancer Center, Newark, Delaware
  - Goergetown-Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Atlantic Melanoma Center, Morristown, New Jersey
  - Duke Cancer Institute, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Omaveloxolone 5 mg & Nivolumab: Omaveloxolone (RTA 408) capsules, 5 mg taken orally once daily for 169 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Omaveloxolone Capsules (2.5 mg/capsule): Capsules containing 2.5 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
  Nivolumab (240 mg): Sterile solution containing nivolumab to be delivered intravenously at 240 mg
- Omaveloxolone 10 mg & Nivolumab: Omaveloxolone (RTA 408) capsules, 10 mg taken orally once daily for 169 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Nivolumab (240 mg): Sterile solution containing nivolumab to be delivered intravenously at 240 mg
  Omaveloxolone Capsules (10 mg/capsule): Capsules containing 10 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
- Omaveloxolone 20 mg & Nivolumab: Omaveloxolone (RTA 408) capsules, 20 mg taken orally once daily for 169 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Nivolumab (240 mg): Sterile solution containing nivolumab to be delivered intravenously at 240 mg
  Omaveloxolone Capsules (10 mg/capsule): Capsules containing 10 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
- Omaveloxolone 100 mg & Nivolumab: Omaveloxolone (RTA 408) capsules, 100 mg taken orally once daily for 169 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Nivolumab (240 mg): Sterile solution containing nivolumab to be delivered intravenously at 240 mg
  Omaveloxolone Capsules (50 mg/capsule): Capsules containing 50 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
- Omaveloxolone 150 mg & Nivolumab: Omaveloxolone (RTA 408) capsules, 150 mg taken orally once daily for 169 weeks, plus nivolumab (240 mg) administered every two weeks as clinically indicated.
  Nivolumab (240 mg): Sterile solution containing nivolumab to be delivered intravenously at 240 mg
  Omaveloxolone Capsules (50 mg/capsule): Capsules containing 50 mg of omaveloxolone per capsule to the dosage indicated in the Arm Label
Period: Overall Study
Arm/Group | Omaveloxolone 5 mg & Ipilimumab | Omaveloxolone 10 mg & Ipilimumab | Omaveloxolone 5 mg & Nivolumab | Omaveloxolone 10 mg & Nivolumab | Omaveloxolone 20 mg & Nivolumab | Omaveloxolone 100 mg & Nivolumab | Omaveloxolone 150 mg & Nivolumab
Started | 6 | 6 | 6 | 6 | 6 | 6 | 5
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 6 | 6 | 6 | 6 | 6 | 6 | 5
Not completed — Adverse Event | 1 | 1 | 2 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 4 | 5 | 4 | 5 | 4 | 5 | 4
Not completed — Sponsor termination of study | 1 | 0 | 0 | 1 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omaveloxolone 5 mg & Ipilimumab | Omaveloxolone 10 mg & Ipilimumab | Omaveloxolone 5 mg & Nivolumab | Omaveloxolone 10 mg & Nivolumab | Omaveloxolone 20 mg & Nivolumab | Omaveloxolone 100 mg & Nivolumab | Omaveloxolone 150 mg & Nivolumab | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.17 (18.713) | 53.5 (8.24) | 68.33 (12.42) | 51.67 (11.29) | 60.5 (13.882) | 65 (7.321) | 65 (5.958) | 60.3 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 0 | 4 | 4 | 1 | 17
  Male | 3 | 4 | 3 | 6 | 2 | 2 | 4 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 6 | 6 | 5 | 5 | 6 | 6 | 5 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 6 | 6 | 6 | 6 | 6 | 6 | 5 | 41
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Measure of Efficacy of the Phase 2 Dose of RTA 408 in Combination With Nivolumab Using Overall Response Rate (ORR; Complete Plus Partial Responses) According to RECIST Version 1.1 Criteria
Description: Best overall response rate (ORR) is defined as the proportion of patients with complete or partial tumor size reduction according to RECIST v1.1 criteria. Stable disease is not a component of ORR.
  Complete response: Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial reduction: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  The first occurrence of a response is considered an unconfirmed response. A CR or PR which persists to the next tumor burden assessment is then considered a confirmed response. Confirmed plus unconfirmed best overall response are presented. A subject may be counted twice if best unconfirmed response and best confirmed response are different.
Time Frame: From enrollment up to the time of disease progression, up to 172 weeks for participants receiving Omaveloxolone in combination with Ipilimumab and 173 weeks for participants receiving Omaveloxolone combination with Nivolumab
Population: Evaluable analysis set (EAS) is defined as all enrolled patients having received at least two weeks of study drug before disease progression and excludes patients who discontinued from study for reasons other than an adverse event prior to first tumor restaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Omaveloxolone 5 mg & Ipilimumab | Omaveloxolone 10 mg & Ipilimumab | Omaveloxolone 5 mg & Nivolumab | Omaveloxolone 10 mg & Nivolumab | Omaveloxolone 20 mg & Nivolumab | Omaveloxolone 100 mg & Nivolumab | Omaveloxolone 150 mg & Nivolumab
Number analyzed (Participants) | 6 | 3 | 6 | 4 | 5 | 5 | 5
Participants
  Best Overall Responses | 6 | 0 | 5 | 2 | 3 | 3 | 4
  Progressive Disease | 3 | 0 | 3 | 0 | 1 | 3 | 2
  Stable Disease | 1 | 0 | 1 | 1 | 1 | 1 | 1
  Partial Response | 3 | 0 | 0 | 2 | 2 | 0 | 2
  Complete Response | 0 | 0 | 1 | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from time of the first dose of study drug up to the time of disease progression, up to 172 weeks for participants receiving Omaveloxolone in combination with Ipilimumab and 173 weeks for participants receiving Omaveloxolone combination with Nivolumab.
Description: Collection of adverse event information was done based on regular investigator assessment during patients visits.
Arm/Group | Omaveloxolone 5 mg & Ipilimumab | Omaveloxolone 10 mg & Ipilimumab | Omaveloxolone 5 mg & Nivolumab | Omaveloxolone 10 mg & Nivolumab | Omaveloxolone 20 mg & Nivolumab | Omaveloxolone 100 mg & Nivolumab | Omaveloxolone 150 mg & Nivolumab
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 1/6 | 1/6 | 2/6 | 0/6 | 1/5
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 1/6 | 3/6 | 2/6 | 2/6 | 2/5
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 6/6 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Omaveloxolone 5 mg & Ipilimumab (N=6) | Omaveloxolone 10 mg & Ipilimumab (N=6) | Omaveloxolone 5 mg & Nivolumab (N=6) | Omaveloxolone 10 mg & Nivolumab (N=6) | Omaveloxolone 20 mg & Nivolumab (N=6) | Omaveloxolone 100 mg & Nivolumab (N=6) | Omaveloxolone 150 mg & Nivolumab (N=5)
Lung Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oesophageal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebral thrombosis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Omaveloxolone 5 mg & Ipilimumab (N=6) | Omaveloxolone 10 mg & Ipilimumab (N=6) | Omaveloxolone 5 mg & Nivolumab (N=6) | Omaveloxolone 10 mg & Nivolumab (N=6) | Omaveloxolone 20 mg & Nivolumab (N=6) | Omaveloxolone 100 mg & Nivolumab (N=6) | Omaveloxolone 150 mg & Nivolumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 2 | 0 | 0 | 1 | 2
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Multiple lentigines syndrome (Congenital, familial and genetic disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophysitis (Endocrine disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye disorder (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mydriasis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vision blurred (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 2 | 2 | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 2 | 3 | 3 | 3 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1 | 1 | 2 | 4 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 2 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucous stools (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 4 | 4 | 1 | 2 | 4 | 0
Oesophageal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 5 | 5 | 1 | 6 | 1 | 3
Gait disturbance (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaise (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nodule (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 2 | 2 | 0 | 0 | 1 | 0
Pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 2 | 1 | 2 | 1 | 1 | 1 | 2
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Clostridial infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Skin infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 1 | 0 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 3 | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Open wound (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 3 | 2 | 2 | 1 | 0 | 1 | 1
Aspartate aminotransferase increased (Investigations) | 3 | 1 | 2 | 0 | 1 | 1 | 1
Biopsy site unspecified abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 2 | 2 | 2 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood corticotrophin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood testosterone decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Cardiac murmur (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2 | 3 | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 2 | 2 | 1 | 0 | 1 | 0
Lymphocyte count increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oesophagogastroduodenoscopy (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 0
Serum ferritin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Very low density lipoprotein increased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2 | 0
Weight decreased (Investigations) | 0 | 2 | 1 | 0 | 0 | 1 | 2
Weight increased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0 | 2 | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 3 | 1 | 2 | 1 | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1 | 1 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Benign vaginal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 1 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 3 | 0 | 3 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 2 | 1 | 3 | 2 | 3 | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Speech disorder developmental (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased activity (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 3 | 1 | 1 | 1 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1 | 3 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 2 | 1 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 1 | 1 | 3
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 2 | 1 | 2 | 0 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 0 | 1 | 0 | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Micrographic skin surgery (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 1 | 1 | 1 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 1 | 1 | 1 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2016-11-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT02259231/Prot_000.pdf
  • Statistical Analysis Plan (2019-10-25): https://cdn.clinicaltrials.gov/large-docs/31/NCT02259231/SAP_001.pdf